CLINICAL TRIAL: NCT04403763
Title: A First-in-Human, Phase 1/2, Dose-ascending, Multicenter, Masked, Randomized, Vehicle-controlled Study Evaluating the Safety, Tolerability, and Pharmacokinetics of AGN-241622 in Healthy Participants and Participants With Presbyopia (Stage 1 and Stage 2) and Efficacy in Participants With Presbyopia (Stage 2)
Brief Title: Phase 1/2 Study of AGN-241622 in Healthy Participants and Participants With Presbyopia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-101-013
Record Dates: First submitted 2020-05-01; First posted 2020-05-27 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Presbyopia
Keywords: Presbyopia,Healthy Subject,Subjects with Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Placebo Dose (Placebo Comparator): Administered as single drop in one or both eyes
  Interventions: Drug: Vehicle
- Cohort 1: AGN-241622 Dose 1 (Low Dose) (Experimental): Administered as single drop in one eye
  Interventions: Drug: AGN-241622
- Cohort 2: AGN-241622 Dose 2 (Medium Dose) (Experimental): Administered as single drop in one eye
  Interventions: Drug: AGN-241622
- Cohort 3: AGN-241622 Dose 3 (High Dose) (Experimental): Administered as single drop in one eye
  Interventions: Drug: AGN-241622
- Cohort 4: AGN-241622 Dose 1 (Low Dose) (Experimental): Administered as a single drop in each eye
  Interventions: Drug: AGN-241622
- Cohort 5: AGN-241622 Dose 2 (Medium Dose) (Experimental): Administered as single drop in each eye
  Interventions: Drug: AGN-241622
- Cohort 6: AGN-241622 Dose 3 (High Dose) (Experimental): Administered as single drop in each eye
  Interventions: Drug: AGN-241622

INTERVENTIONS:
Drug: AGN-241622 — Topical eye drop
  Arms: Cohort 1: AGN-241622 Dose 1 (Low Dose); Cohort 2: AGN-241622 Dose 2 (Medium Dose); Cohort 3: AGN-241622 Dose 3 (High Dose); Cohort 4: AGN-241622 Dose 1 (Low Dose); Cohort 5: AGN-241622 Dose 2 (Medium Dose); Cohort 6: AGN-241622 Dose 3 (High Dose)
Drug: Vehicle — Topical eye drop
  Arms: Placebo Dose

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AGN-241622 ophthalmic solution for the first time in human participants

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 65 at the time of study participation.
* Be a nonsmoker and nonuser of nicotine-containing products within the previous 1 year.
* Be able and willing to follow study instructions and complete all required study visits in the opinion of the study doctor.

Exclusion Criteria:

* History of alcohol or substance abuse within the 5 years prior to study participation.
* Enrollment in another investigational drug or device study within 30 days of study participation.
* Women who are pregnant, nursing, or planning a pregnancy during the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - United Medical Research Institute /ID# 234612, Inglewood, California
  - Global Research Foundation /ID# 237353, Los Angeles, California
  - North Valley Eye Medical Group, Inc. /ID# 236686, Mission Hills, California
  - The Eye Research Foundation /ID# 234526, Newport Beach, California
  - Quantum Clinical Trials /ID# 237330, Miami Beach, Florida
  - Kannarr Eye Care /ID# 236718, Pittsburg, Kansas
  - The Eye Care Institute /ID# 234507, Louisville, Kentucky
  - Total Eye Care, PA /ID# 234454, Memphis, Tennessee
  - PPD Clinical Research Unit - Austin /ID# 237644, Austin, Texas
  - Eye associates /ID# 236502, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance — http://www.AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was to be conducted in 3 stages (Stage 1, Stage 2a, and Stage 2b) with participants being randomized to different stages with dose cohorts based on criteria. Due to Sponsor decision, the study was terminated before completion. This decision was not taken due to any safety reasons.
Groups:
- Placebo Dose: Administered as a single drop in one or both eyes
  Vehicle: Topical eye drop
Period: Stage 1
Arm/Group | Placebo Dose | Cohort 1: AGN-241622 Dose 1 (Low Dose) | Cohort 2: AGN-241622 Dose 2 (Medium Dose) | Cohort 3: AGN-241622 Dose 3 (High Dose) | Cohort 4: AGN-241622 Dose 1 (Low Dose) | Cohort 5: AGN-241622 Dose 2 (Medium Dose) | Cohort 6: AGN-241622 Dose 3 (High Dose)
Started | 10 | 9 | 10 | 9 | 0 | 0 | 0
Completed | 9 | 8 | 9 | 9 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Participant did not dose due to Sponsor decision | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Early termination due to PK tube failure | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Stage 2A
Arm/Group | Placebo Dose | Cohort 1: AGN-241622 Dose 1 (Low Dose) | Cohort 2: AGN-241622 Dose 2 (Medium Dose) | Cohort 3: AGN-241622 Dose 3 (High Dose) | Cohort 4: AGN-241622 Dose 1 (Low Dose) | Cohort 5: AGN-241622 Dose 2 (Medium Dose) | Cohort 6: AGN-241622 Dose 3 (High Dose)
Started | 9 | 0 | 0 | 0 | 12 | 11 | 10
Completed | 9 | 0 | 0 | 0 | 12 | 11 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consists of all randomized participants.
Groups:
- Cohort 5: AGN-241622 Dose 2 (Medium Dose); Cohort 6: AGN-241622 Dose 3 (High Dose): Administered as a single drop in each eye
  AGN-241622: Topical eye drop
- Total: Total of all reporting groups
Arm/Group | Placebo Dose | Cohort 1: AGN-241622 Dose 1 (Low Dose) | Cohort 2: AGN-241622 Dose 2 (Medium Dose) | Cohort 3: AGN-241622 Dose 3 (High Dose) | Cohort 4: AGN-241622 Dose 1 (Low Dose) | Cohort 5: AGN-241622 Dose 2 (Medium Dose) | Cohort 6: AGN-241622 Dose 3 (High Dose) | Total
Number analyzed (Participants) | 19 | 9 | 10 | 9 | 12 | 11 | 10 | 80
Age, Customized [Count of Participants; unit: Participants]
  <=50 | 8 | 6 | 2 | 2 | 2 | 6 | 1 | 27
  >50 | 11 | 3 | 8 | 7 | 10 | 5 | 9 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 8 | 3 | 7 | 9 | 5 | 52
  Male | 5 | 3 | 2 | 6 | 5 | 2 | 5 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 1 | 1 | 2 | 5 | 0 | 20
  Not Hispanic or Latino | 14 | 3 | 9 | 8 | 10 | 6 | 10 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 0 | 2 | 4 | 2 | 0 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 2 | 0 | 4 | 1 | 4 | 16
  White | 10 | 8 | 6 | 5 | 6 | 10 | 5 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Number of Participants Experiencing a Treatment Emergent Adverse Event After Single Administration of AGN-241622
Description: The number of participants who experience one or more TEAE during the treatment period
Time Frame: Up to 2 days
Population: The safety population consists of all participants who received at least 1 administration of study intervention. Participants will be summarized according to the study intervention they actually received.
Measure: Number; unit: participants
Groups:
- Stage 1 Placebo Dose: Administered as single drop in one eye
  Vehicle: Topical eye drop
Arm/Group | Stage 1 Placebo Dose | Cohort 1: AGN-241622 Dose 1 (Low Dose) | Cohort 2: AGN-241622 Dose 2 (Medium Dose) | Cohort 3: AGN-241622 Dose 3 (High Dose)
Number analyzed (Participants) | 9 | 8 | 9 | 9
participants
  Ocular | 1 | 7 | 1 | 0
  Non-ocular | 2 | 1 | 3 | 0

2. Primary Outcome: Stage 2a: Number of Patients Experiencing a Treatment Emergent Adverse Event After Repeat Administration of AGN-241622
Description: The number of patients who experience one or more TEAE during the treatment period
Time Frame: 14 Days
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Stage 2a Placebo Dose: Administered as single drop in each eye
  Vehicle: Topical eye drop
Arm/Group | Stage 2a Placebo Dose | Cohort 4: AGN-241622 Dose 1 (Low Dose) | Cohort 5: AGN-241622 Dose 2 (Medium Dose) | Cohort 6: AGN-241622 Dose 3 (High Dose)
Number analyzed (Participants) | 9 | 12 | 11 | 10
participants
  Ocular | 1 | 0 | 2 | 1
  Non-ocular | 0 | 0 | 1 | 1

3. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Terminal Elimination Half-life (T1/2) of AGN-241622
Description: To evaluate the systemic and local pharmacokinetics of AGN-241622 administered once unilaterally in healthy participants
Time Frame: Day 1
Reporting Status: Not Posted

4. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Terminal Elimination Rate Constant (λz) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

5. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Maximum Plasma Concentrations (Cmax) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

6. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Time of Maximum Plasma Concentrations (Tmax) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

7. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Apparent Total Clearance of AGN-241622 From Plasma (CL/F)
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

8. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Volume of Distribution During the Terminal Elimination Phase (Vz/F) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

9. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to Time t (AUC0-t) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

10. Secondary Outcome: Stage 1 Plasma Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

11. Secondary Outcome: Stage 1 Tears Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to Time t (AUC0-t) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

12. Secondary Outcome: Stage 1 Tears Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

13. Secondary Outcome: Stage 1 Tears Pharmacokinetics: Maximum Plasma Concentrations (Cmax) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

14. Secondary Outcome: Stage 1 Tears Pharmacokinetics: Time of Maximum Plasma Concentrations (Tmax) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

15. Secondary Outcome: Stage 1 Tears Pharmacokinetics: Terminal Elimination Rate Constant (λz) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

16. Secondary Outcome: Stage 1 Tears Pharmacokinetics: Terminal Elimination Half-life (T1/2) of AGN-241622
Description: as for outcome 3
Time Frame: Day 1
Reporting Status: Not Posted

17. Secondary Outcome: Stage 1: Pupil Diameter Measurement
Description: To evaluate the target receptor engagement of AGN-241622 as compared with vehicle administered once, unilaterally in healthy participants
Time Frame: Day 1
Reporting Status: Not Posted

18. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to Time t (AUC0-t) of AGN-241622
Description: To evaluate the systemic and local pharmacokinetics of AGN-241622 after repeat bilateral administration in participants with presbyopia
Time Frame: 14 Days
Reporting Status: Not Posted

19. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Area Under the Plasma/Tear Concentration Versus Time Curve From Time 0 to the End of the Dosing Period (AUC0-tau) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

20. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Maximum Plasma Concentrations (Cmax) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

21. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Minimum Plasma Concentrations (Cmin) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

22. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Time of Maximum Plasma Concentrations (Tmax) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

23. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Terminal Elimination Rate Constant (λz) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

24. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Terminal Elimination Half-life (T1/2) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

25. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Apparent Total Clearance of AGN-241622 From Plasma (CL/F)
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

26. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Volume of Distribution During the Terminal Elimination Phase (Vz/F) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

27. Secondary Outcome: Stage 2a Plasma Pharmacokinetics: Accumulation Ratio of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

28. Secondary Outcome: Stage 2a Tears Pharmacokinetics: Area Under the Concentration-time Curve From Time 0 to Time t (AUC0-t) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

29. Secondary Outcome: Stage 2a Tears Pharmacokinetics: Area Under the Plasma/Tear Concentration Versus Time Curve From Time 0 to the End of the Dosing Period (AUC0-tau) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

30. Secondary Outcome: Stage 2a Tears Pharmacokinetics: Maximum Plasma Concentrations (Cmax) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

31. Secondary Outcome: Stage 2a Tears Pharmacokinetics: Time of Maximum Plasma Concentrations (Tmax) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

32. Secondary Outcome: Stage 2a Tears Pharmacokinetics: Terminal Elimination Rate Constant (λz) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

33. Secondary Outcome: Stage 2a Tears Pharmacokinetics: Terminal Elimination Half-life (T1/2) of AGN-241622
Description: as for outcome 18
Time Frame: 14 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 Weeks
Groups:
- Cohort 1: AGN-241622 Dose 1; Cohort 2: AGN-241622 Dose 2; Cohort 3: AGN-241622 Dose 3: Administered as single drop in one eye
  AGN-241622: Topical eye drop
- Cohort 4: AGN-241622 Dose 1; Cohort 5: AGN-241622 Dose 2; Cohort 6: AGN-241622 Dose 3: Administered as a single drop in each eye
  AGN-241622: Topical eye drop
Arm/Group | Stage 1 Placebo Dose | Cohort 1: AGN-241622 Dose 1 | Cohort 2: AGN-241622 Dose 2 | Cohort 3: AGN-241622 Dose 3 | Stage 2a Placebo Dose | Cohort 4: AGN-241622 Dose 1 | Cohort 5: AGN-241622 Dose 2 | Cohort 6: AGN-241622 Dose 3
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/9 | 0/9 | 0/12 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/9 | 0/9 | 0/12 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 3/9 | 7/8 | 4/9 | 0/9 | 1/9 | 0/12 | 3/11 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Stage 1 Placebo Dose (N=9) | Cohort 1: AGN-241622 Dose 1 (N=8) | Cohort 2: AGN-241622 Dose 2 (N=9) | Cohort 3: AGN-241622 Dose 3 (N=9) | Stage 2a Placebo Dose (N=9) | Cohort 4: AGN-241622 Dose 1 (N=12) | Cohort 5: AGN-241622 Dose 2 (N=11) | Cohort 6: AGN-241622 Dose 3 (N=10)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
EYE IRRITATION (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
EYE PRURITUS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
PUNCTATE KERATITIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0/9 (0) | 2 (3) | 1 (2)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 1 (1) | 0 (0)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
BLOOD PRESSURE DIASTOLIC INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
PROTEIN URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/9 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT04403763/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT04403763/SAP_003.pdf